CLINICAL TRIAL: NCT04279509
Title: Selecting Chemotherapy With High-throughput Drug Screen Assay Using Patient Derived Organoids in Patients With Refractory Solid Tumours (SCORE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC01/01/19
Record Dates: First submitted 2020-02-10; First posted 2020-02-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Organoids; HNSCC; Epithelial Ovarian Cancer; Colorectal Cancer
Keywords: Organoid
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Ovarian Epithelial; Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patient (Experimental): Histological or cytological diagnosis of head and neck squamous cell carcinoma (HNSCC), colorectal, breast or epithelial ovarian cancer.
  Interventions: Procedure: Tumor Core Biopsy; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Tumor Core Biopsy — Performed up to a maximum of 3 time points - baseline upon study enrolment, at the completion of treatment, and upon disease progression.
  Four to six tumour core samples will be obtained at each time point. At least two tumour cores will be sent fresh to Invitrocue Pte Ltd for generation of patient-derived organoids for drug-panel screening, at least 1-2 tumour cores at each time point will be stored in formalin and paraffin-embedded for immunohistochemistry analysis of biomarkers, while the remaining 1-2 tumour cores will be stored in liquid nitrogen for subsequent DNA, RNA and protein extraction for biomarker studies including gene expression and proteomics analyses.
Procedure: Blood sampling — Germline DNA at baseline for pharmacogenetics analysis. Serial plasma samples for circulating tumour cells and biomarkers, at baseline, prior to day 1 of each cycle while on treatment, at the end of treatment (either upon disease progression or upon completion of predetermined cycles of chemotherapy).

SUMMARY:
This is a single-centre study based on the Simon 2-stage optimax design: 12 patients will be enrolled initially (Stage I), which will then be expanded to a further 13 patients (Stage II) if 3 or more patients enrolled in stage I of the study achieve an objective response with the chemotherapeutic agent selected by the drug screen assay. A total of 25 patients will be included in both stages of study.

Patients enrolled on study will undergo a fresh biopsy of tumour lesion to obtain cells that will be used to generate patient-derived tumour organoids based on the Invitrocue technology. Organoids will then be subjected to a 10-drug panel screening including: 5-fluorouracil, carboplatin, cyclophosphamide, docetaxel, doxorubicin, gemcitabine, irinotecan, oxaliplatin, paclitaxel and vinorelbine. A further 5 drugs (etoposide, ifosfamide, methotrexate, pemetrexed and topotecan) will be screened if sufficient organoids are grown from the biopsy samples within the screening period.

Physicians will be informed of the results, and choice of chemotherapy will be based on an IRS score of 70% or above. If more than 1 candidate drug with IRS of 70% or above is identified, the physician will exercise his/her discretion to select the most suitable drug based on patient's comorbidities and organ function.

DETAILED DESCRIPTION:
Investigators hypothesize that high-throughput screening on patient-derived tumour organoids can be used as an adjunct tool to aid treatment selection in patients with cancer. Using the IRS, drugs with high IRS (defined as a score of 70% and above) will have a high probability of inducing objective response (either a complete or partial response by RECIST criteria) in patients with refractory cancers. Conversely, IRS of drugs for which the patients have been treated and experienced clinical progression on will be low (defined as a score of 50% or below).

Primary Objectives

-To prospectively determine if a high-throughput drug screen assay using patient tumour-derived organoids can accurately select a chemotherapeutic agent that results in objective response in patients with refractory solid tumours

Secondary Objectives

* To assess the IRS measured on tumour-derived organoid drug screen assay of chemotherapeutic agents to which patients had previously progressed on clinically
* To assess changes in IRS pre and post-chemotherapy treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years.
* Histological or cytological diagnosis of head and neck squamous cell carcinoma (HNSCC), colorectal, breast or epithelial ovarian cancer.
* ECOG 0-1.
* At least 1 tumour lesion (primary or metastatic) amenable to fresh biopsy
* At least 1 measurable tumour lesions based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Has documented progressive disease from last line of therapy.
* Able to wait at least 4 to 6 weeks before initiating the next line of anti-cancer therapy.
* Has received at least 2 line of palliative systemic therapy:

  (i) Breast cancer: must have received prior anthracyclines and taxanes in the neoadjuvant, adjuvant or palliative setting, unless either of these drugs were contraindicated due to organ dysfunction and/or comorbidities (ii) Ovarian cancer: must have received prior taxanes and platinums in the neoadjuvant, adjuvant or palliative setting (iii)HNSCC: must have received prior platinums, taxanes, and 5-fluorouracil in the neoadjuvant, adjuvant or palliative setting (iv)Colorectal cancer: must have received prior 5-fluorouracil, oxaliplatin and irinotecan in the neoadjuvant, adjuvant or palliative setting
* Adequate organ function including the following:

  (i)Bone marrow:
  * Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥100 x 109/L
  * Hemoglobin ≥ 8 x 109/L

(ii) Hepatic:

* Bilirubin ≤ 1.5 x upper limit of normal (ULN),
* ALT or AST ≤ 2.5x ULN,(or ≤ 5X with liver metastases)

(iii) Renal:

◦Creatinine ≤ 1.5x ULN

* Signed informed consent from patient or legal representative.
* Able to comply with study-related procedures.

Exclusion Criteria:

* Pace of cancer progression requiring commencement of anti-cancer therapy within 4 to 6 weeks.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Overall radiological response rate | 2 years
  Measured by RECIST of the entire study cohort
Correlation between patient genotype, tumor biomarkers and blood biomarkers with clinical outcome | 2 years
  Clinical Outcome include Radiological response, progression-free survival, grade 3-4 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniel VC, Marchionni L, Hierman JS, Rhodes JT, Devereux WL, Rudin CM, Yung R, Parmigiani G, Dorsch M, Peacock CD, Watkins DN. A primary xenograft model of small-cell lung cancer reveals irreversible changes in gene expression imposed by culture in vitro. Cancer Res. 2009 Apr 15;69(8):3364-73. doi: 10.1158/0008-5472.CAN-08-4210. Epub 2009 Apr 7. PMID 19351829
- [Result] Jones S, Anagnostou V, Lytle K, Parpart-Li S, Nesselbush M, Riley DR, Shukla M, Chesnick B, Kadan M, Papp E, Galens KG, Murphy D, Zhang T, Kann L, Sausen M, Angiuoli SV, Diaz LA Jr, Velculescu VE. Personalized genomic analyses for cancer mutation discovery and interpretation. Sci Transl Med. 2015 Apr 15;7(283):283ra53. doi: 10.1126/scitranslmed.aaa7161. PMID 25877891